CLINICAL TRIAL: NCT01888991
Title: Substrate Oxidation Does Not Affect Short Term Food Intake in Healthy Boys and Men.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIHR kids_26570; CIHR MOP-111250 (Other Grant/Funding Number: 111250)
Record Dates: First submitted 2013-06-22; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Food Intake Regulation; Substrate Oxidation
Keywords: Glucose; Exercise; Metabolic flexibility; Substrate Oxidation; Food intake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- water with resting condition (No Intervention)
- glucose with resting condition (Experimental)
  Interventions: Other: Glucose Preload and Exercise Intervention
- water with exercise condition (Experimental)
  Interventions: Other: Glucose Preload and Exercise Intervention
- glucose with exercise condition (Experimental)
  Interventions: Other: Glucose Preload and Exercise Intervention

INTERVENTIONS:
Other: Glucose Preload and Exercise Intervention — A glucose preload and exercise were administered to examine the modulate substrate oxidation
  Arms: glucose with exercise condition; glucose with resting condition; water with exercise condition

SUMMARY:
The purpose of this study is to investigate the effect of substrate oxidation, expressed by RER, on food intake regulation and net energy balance.

DETAILED DESCRIPTION:
The relationship between substrate oxidation as measured by respiratory exchange ratio (RER) and food intake is undefined. This study is examining the effects of three modulators of substrate oxidation (RER), a glucose preload, exercise and age food intake regulation and net energy balance in normal-weight boys (9-12 y) and men (20-30 y).

Subjects (15 boys, 15 men) were measured in random order with treatments of beverages of either water or glucose followed by either moderate exercise or rest for 40 min. Measures included RER via indirect calorimetry, energy expenditure, subjective appetite, food intake measured at an ad libitum pizza meal and net energy balance as the sum of the calories of the glucose preload + calories from the pizza lunch minus energy expended at exercise or rest.

ELIGIBILITY:
Inclusion Criteria:

* Born at full term
* Men Age:20-29 years/BMI: 20-25
* Boys Age 9-11/BMI percentile: 15th to 85th:

Exclusion Criteria:

* Smokers
* Dieters
* Individuals with lactose intolerance, allergies to milk and dairy products
* Individuals with gastrointestinal problems
* Individuals with diabetes or other metabolic diseases
* Individuals scoring ≥ 11 on an Eating Habit Questionnaire

Ages: 9 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Food Intake | 60 - 90 min in the study
  Energy intake from the ad libitum the pizza meal at 60 min was calculated based on the weight consumed and the compositional information provided by the manufacturer.

SECONDARY OUTCOMES:
Net Energy Balance | 0-90 min in the study
  Will be calculated from the energy consumed by the glucose preload and the pizza meal minus energy expended at the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tamam S, Bellissimo N, Patel BP, Thomas SG, Anderson GH. Overweight and obese boys reduce food intake in response to a glucose drink but fail to increase intake in response to exercise of short duration. Appl Physiol Nutr Metab. 2012 Jun;37(3):520-9. doi: 10.1139/h2012-038. Epub 2012 Apr 25. PMID 22530879
- [Background] Bellissimo N, Thomas SG, Goode RC, Anderson GH. Effect of short-duration physical activity and ventilation threshold on subjective appetite and short-term energy intake in boys. Appetite. 2007 Nov;49(3):644-51. doi: 10.1016/j.appet.2007.04.004. Epub 2007 Apr 22. PMID 17537539
- [Background] Bozinovski NC, Bellissimo N, Thomas SG, Pencharz PB, Goode RC, Anderson GH. The effect of duration of exercise at the ventilation threshold on subjective appetite and short-term food intake in 9 to 14 year old boys and girls. Int J Behav Nutr Phys Act. 2009 Oct 9;6:66. doi: 10.1186/1479-5868-6-66. PMID 19818131
- [Derived] Hunschede S, El Khoury D, Antoine-Jonville S, Smith C, Thomas S, Anderson GH. Acute changes in substrate oxidation do not affect short-term food intake in healthy boys and men. Appl Physiol Nutr Metab. 2015 Feb;40(2):168-77. doi: 10.1139/apnm-2014-0188. Epub 2014 Oct 22. PMID 25603432